CLINICAL TRIAL: NCT00521482
Title: Intensive Dose Temozolomide Treatment or Temozolomide With Thalidomide Treatment in Recurrent Glioblastoma After Standard Therapy:a Randomized Phase II Trial
Brief Title: Temozolomide vs. Temozolomide and Thalidomide Treatment in Recurrent Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMZ/05; P04932
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2007-08-28 (Estimated); Status verified 2007-08

CONDITIONS: Glioblastoma
Keywords: recurrent; after standard therapy
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Temozolomide; Thalidomide; Myrin P

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Temozolomide 75 mg/m2 daily for 21 days during each 28-day cycle until tumor progression.
  Interventions: Drug: Temozolomide
- B (Experimental): Temozolomide 200 mg/m2 for 5 days during each 28-day cycle plus Thalidomide 100 mg for 2 weeks, thereafter 200 mg daily continuously until tumor progression.
  Interventions: Drug: Temozolomide plus Thalidomide

INTERVENTIONS:
Drug: Temozolomide
  Other Names: Temodal
  Arms: A
Drug: Temozolomide plus Thalidomide
  Other Names: Temodal; plus; Myrin
  Arms: B

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of intensive dose temozolomide treatment alone in parallel to a combination with thalidomide in patients with recurrent glioblastoma after standard therapy.

In the treatment arm A of the study it will be investigated whether or not continuous dosing of temozolomide may overcome alkylator resistance in patients with glioblastoma who progress on the 5/28 day dosing regimen.

For treatment arm B it is postulated that the combination of thalidomide and temozolomide is effective with respect to time to progression and progression-free survival due to the fact that temozolomide and thalidomide have different mechanisms of action.

DETAILED DESCRIPTION:
* Primary objectives: To determine the proportion of patients with progression- free survival after 6 months of intensive dose temozolomide treatment alone or in combination with thalidomide in patients with recurrent glioblastoma multiforme after standard therapy.
* Secondary objectives: To assess the effects on tumor growth. To determine the time to disease progression. To determine the proportion of patients with progression- free survival. To assess the safety of intensive dose temozolomide treatment alone or in combination with thalidomide.
* Explorative evaluations: To assess health related Quality of Life. To assess cognitive functioning. To compare the two treatment arms in terms of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 to 70 years
2. Histologically proven glioblastoma, WHO grade IV
3. Evidence of tumor recurrence or progression by MRI at least 3 months after radiation treatment
4. Prior radiation treatment with 60 Gy in 2-Gy fractions; concurrent daily temozolomide 75 mg/m2 daily for 42 days (max. 49 days); adjuvant temozolomide 150 - 200mg/m2 for 5 days during each 28-day cycle (max. 6 cycles)
5. Patient should have received a minimum of 2 cycles of adjuvant chemotherapy with temozolomide after concomitant regime of temozolomide and Radiotherapy
6. Patient had recovered from the effects of surgery
7. Karnofsky Performance Status of ≥70
8. Mini-Mental State Examination score >25
9. Adequate hepatic function: AST <52 U/l, ALT <50 U/l, AP ≤129 U/l
10. Adequate hematological values: neutrophils ≥1.5 x 109/l, thrombocytes ≥100 x 109/l
11. Adequate renal function: clearance <110 μmol/l
12. Written informed consent before entering the study

Exclusion Criteria:

1. Other severe underlying diseases
2. Significant renal, hepatic or bone marrow impairment
3. Pregnant women, women who are breast feeding, and women of childbearing potential who are not using chemical or mechanical contraception (prescription oral contraceptives, abstinence, condoms with spermicide, surgical sterilization, diaphragm with spermicide, or intrauterine device) or have a positive pregnancy test
4. Known Acquired Immune Deficiency Syndrome (AIDS)
5. Known hypersensitivity to temozolomide, dacarbazine or thalidomide (or any of the excipients)
6. Any concomitant drugs contraindicated for use with temozolomide (according to the product information in the Swiss drug compendium) and thalidomide (investigator's brochure, international product information).
7. Concurrent treatment with other experimental drugs or other anti-cancer therapy; treatment within a clinical trial within 30 days prior to trial entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-09; Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with progression free survival | 6 months

SECONDARY OUTCOMES:
Proportion of patients with a clinical response. Time to disease progression. Progression free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Miroslava Bjeljac, MD, Principal Investigator — University of Zurich
Locations (1):
- University Zurich, Departement of Neurosurgery, Zurich, Switzerland